CLINICAL TRIAL: NCT02711319
Title: Non-invasive Brain Stimulation in SCI
Brief Title: Non-invasive Brain Stimulation for Gait Improvement in Patients With Spinal Cord Injury
Acronym: SCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Guttmann (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Joan Vidal, MD, PhD, Institut Guttmann
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI10/00442
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Functional Improvement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (real) rTMS (ACTIVE GROUP) (Active Comparator): The patients were randomly distributed in two study groups: real or sham rTMS group.
  For real rTMS, we applied 2 seconds duration bursts of 20 Hz (40 pulses/burst) with intertrain intervals of 28 seconds, for a total of 1800 pulses over 20 minutes.
  Interventions: Device: rTMS
- sham rTMS (SHAM GROUP) (Sham Comparator): For sham rTMS, the double cone coil was again held over the vertex, but it was disconnected from the main stimulator unit. Instead, a second coil (8-shaped) was connected to the MagStim stimulator, and discharged under the patient's pillow (2).
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: rTMS — For real (active) rTMS, we applied 2 seconds duration bursts of 20 Hz (40 pulses/burst) with intertrain intervals of 28 seconds, for a total of 1800 pulses over 20 minutes
  Other Names: active rTMS; active group; real rTMS
  Arms: active (real) rTMS (ACTIVE GROUP)
Device: sham rTMS — Sham Comparator: sham rTMS (SHAM GROUP)
  For sham rTMS, the double cone coil was again held over the vertex, but it was disconnected from the main stimulator unit. Instead, a second coil (8-shaped) was connected to the MagStim stimulator, and discharged under the patient's pillow (2).
  Other Names: sham group; placebo group
  Arms: sham rTMS (SHAM GROUP)

SUMMARY:
to optimize the functional outcome in early phase of gait rehabilitation in subacute incomplete SCI patients using rTMS as an additional treatment to physical therapy (e.g. to gait training in Lokomat®). Using this add-on therapeutic strategy, we expected larger improvement of gait function than with physical therapy alone.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive and painless procedure to modulate cortical excitability of motor areas and induce changes over the descending corticospinal output. This modulation may be useful to promote active recovery of motor function and to obtain functional benefit from gait rehabilitation. Through the use of repetitive high-frequency rTMS, improvement has been reported in motor and sensory functions measured by American Spinal Cord Injury Association (ASIA) Impairment Scale (AIS), and time to complete a peg-board task in four chronic incomplete cervical SCI patients.

Physical therapy aims to improve function of both undamaged and also, as far as possible, damaged neuronal structures. However, 'reorganization' of neuronal circuits is the target of specific training approaches. Therefore, the challenge is to guide CNS plasticity in order to optimize the functional outcome for a given individual. Hypothesized was that high-frequency rTMS coupled with gait training can improve motor recovery in the lower extremities and locomotion in incomplete SCI patients to a greater degree than sham stimulation.

ELIGIBILITY:
inclusion criteria:

1. had subacute motor incomplete SCI (AIS-C or D),
2. candidate for gait rehabilitation with Lokomat® after cervical or thoracic SCI;
3. stable medical treatment at least one week before and during the study;
4. without limitation of passive range of movement in joints
5. agreed to participate after signing a written informed consent form.

exclusion criteria:

1. unstable clinical state
2. severe spasticity (MAS>=3)
3. disagreed to sign consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ten-meters walking test (10MWT=Time in seconds to walk 10 meters.) | Change from Baseline 10MWT at 4 and 8 weeks
  Patients with or without orthesis were asked to walk at their fastest but most comfortable speed and step length and cadence assessed during the 10MWT (We added the number of steps taken in 10 m. Step length (meters)=distance (m) x 2 / number of stops (heel to heel of same foot). Cadence (steps/min.)=number of steps x 60 / time (seconds))

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Change from Baseline MAS at 4 weeks
  Tests resistance to passive movement about a joint with varying degrees of velocity at knees
--Total motor score from upper (UEMS) and lower extremities (LEMS) | Change from Baseline 1UEMS and LEMS at 4 and 8 weeks
  Total motor score from upper (UEMS) (score 50points) and lower extremities (LEMS) (score 50points) obtained from the standardized AIS clinical exam (total score=100)
Walking Index for SCI (WISCI) II | Change from Baseline WISCI-II at 4 and 8 weeks
  The ranking of severity of gait is based on the severity of the impairment and not on functional independence in the environment.

IPD SHARING:
Plan to Share IPD: Undecided